CLINICAL TRIAL: NCT02340533
Title: The Diagnostic Accuracy of Hysteroscopic Endomyometrial Biopsy in Adenomyosis
Brief Title: Histopathological Diagnosis of Adenomyosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Dina Mohamed Refaat Dakhly, lecturer of obstetrics and gynecology, Woman's Health University Hospital, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: AD0152015
Record Dates: First submitted 2015-01-09; First posted 2015-01-16 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Adenomyosis
Keywords: adenomyosis
MeSH Terms: conditions — Adenomyosis | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- adenomyosis (Experimental): females attending the gynecology outpatient clinic complaining of chronic pelvic congestion will get enrolled in the study. Two dimensional ultrasonography will be performed to asses the presence or absence of adenomyosis or any associated lesions. All the patients were then be subjected to office hysteroscopy and endo-myometrial biopsies will be taken. Histopathological examination of the samples will then be done. From these recruited patients, some will be indicated to perform hysterectomy. The final diagnosis will then be based on the histopathological examination of the specimen retrieved from hysterectomy. The accuracy of the ultrasound and the hysteroscopic endo-myometrial biopsy will then be compared and assessed.
  Interventions: Procedure: hysteroscopic endo-myometrial biopsy; Device: ultrasound

INTERVENTIONS:
Procedure: hysteroscopic endo-myometrial biopsy
Device: ultrasound — two dimensional trans-vaginal ultrasonography

SUMMARY:
The purpose of this study is to develop and evaluate a hysteroscopic endo-myometrial biopsy for diagnosing adenomyosis.

ELIGIBILITY:
Inclusion Criteria:

* females complaining of pelvic congestion: dysmenorrhea, dyspareunia, chronic pelvic pain, menorrhagia, metrorrhagia

Exclusion Criteria:

* refusal of the patient to get enrolled in the study

Ages: 38 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with diagnosis of adenomyosis cases | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dina M Dakhly, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr el aini hospital, Cairo, Cairo Governorate, Egypt